CLINICAL TRIAL: NCT03774277
Title: Chickasaw Healthy Eating Environments Research Study
Acronym: CHEERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Collaborators: The Chickasaw Nation (Unknown); Washington State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7614
Record Dates: First submitted 2018-12-07; First posted 2018-12-12 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Blood Pressure; Body Weight
Keywords: Hypertension; Blood Pressure; DASH-Diet; BMI; American Indian; Food Environment; CBPR; CHEERS; Native American
MeSH Terms: conditions — Body Weight; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Communities (Experimental): Packed Promise for a Healthy Heart intervention, free Tribal Wellness Center membership, a Fitbit, and the AYA culturally based mobile walking app.
  Interventions: Behavioral: Packed Promise for a Healthy Heart
- Control Communities (No Intervention): Free Tribal Wellness Center membership, Fitbit, and the AYA culturally based mobile walking app

INTERVENTIONS:
Behavioral: Packed Promise for a Healthy Heart — Voucher for fresh vegetables and fruits (referred to as a "fresh check"); Home delivered food boxes that contain Dietary Approaches to Stop Hypertension (DASH)-approved ingredients for preparing low-salt, and traditional healthy Chickasaw meals; Heart-healthy recipes (available at getfreshcooking.com) that are tailored to traditional Chickasaw diet and culture; Educational materials; Personalized invitation to attend local cooking demonstrations; Assistance to link the Fitbit and AYA app
  Arms: Intervention Communities

SUMMARY:
This study, the Chickasaw Healthy Eating Environments Research Study (CHEERS), will be conducted in partnership with Chickasaw Nation. CHEERS comprises several mutually reinforcing strategies to improve blood pressure (BP) control in people with hypertension. Environmental strategies include the investigator's innovative "Packed Promise for a Healthy Heart" program that provides hypertensive adults ages 18 and older with a voucher for fresh vegetables and fruits (referred to as a "fresh check") and home delivered food boxes that contain Dietary Approaches to Stop Hypertension (DASH)-approved ingredients for preparing low-salt, and traditional healthy Chickasaw meals. The study facilitates demonstrations of healthy cooking practices in participating communities. At the individual level, tribal members with uncontrolled hypertension will receive heart-healthy recipes (available at getfreshcooking.com) that are tailored to traditional Chickasaw diet and culture, educational materials, along with invitations to attend cooking demonstrations, fresh checks to improve access to fresh produce, and a Chickasaw Nation culturally-informed smartphone walking app called "AYA." At the policy level, CHEERS will culminate in a multimedia documentary presentation for tribal leadership detailing the intervention and featuring personal success stories by hypertensive community members. Study findings, including a health economics assessment, will be used to encourage policies for further expansion of the Packed Promise for a Healthy Heart Program; and policies promoting expansion of brick and mortar grocery outlets in rural Chickasaw communities.

DETAILED DESCRIPTION:
This study is guided by the principles of community-based participatory research (CBPR).

Aims and Methods: Co-led by an AI (Choctaw) Investigator, the study will:

Aim #1: Evaluate CHEERS' ability to improve healthy food access by collecting quantitative data on changes in perceived ability to purchase and prepare healthy food, and by using qualitative methods to evaluate the reach, saturation, and acceptability of the CHEERS intervention.

Aim #2: Measure the intervention's effect on change in BP and secondary outcomes among hypertensive community members with poorly controlled hypertension.

Aim #3: Disseminate a multimedia documentary of the study's findings and evaluate the documentary's effect on tribal leaders across the Chickasaw Nation and other tribal communities.

Innovation: This study will evaluate the effects of a multilevel, tribally-run, food environment intervention. The study will also be one of the few food environment interventions ever implemented in an AI community, and the first to objectively measure its effects on BP and BMI.

Significance and Impact: Study findings, including a health economics assessment, will be used to encourage policies for further expansion of the Packed Promise for a Healthy Heart Program; and policies promoting expansion of brick and mortar grocery outlets in rural Chickasaw communities.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Self-identify as American Indian/Alaska Native
* Currently reside in the four communities and do not plan on moving for 12 months
* Not currently pregnant, or ≥ 6 weeks postpartum
* Ability to understand written and spoken English
* Ability and willingness to follow study protocols
* Self-reported previous diagnosis of hypertension by a medical professional and a measured systolic BP ≥ 130 mm Hg at time of enrollment or no previous hypertension diagnosis and a measured systolic BP ≥ 130 mm Hg at both the initial screening and prior to finalizing enrollment (i.e. on two separate days)

Exclusion Criteria:

- Anyone not meeting the aforementioned inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure | Measured before and after the 6 month intervention
  Targeted 2.9 mm Hg decrease in systolic blood pressure

SECONDARY OUTCOMES:
Food security | Measured before and after the 6 month intervention
  USDA Household Food Security Scale (6 Item Short Module) - The sum of affirmative responses provides a household raw score. Food security status of households with raw scores of 0-1 are high or marginally food secure, raw scores of 2-4 are low secure, and raw scores of 5-6 are very low food secure. High raw scores indicate food insecure households.
Diet | Measured before and after the 6 month intervention
  ASA24, a self-administered recall system (https://asa24.nci.nih.gov/)
Change in body mass index | Measured before and after the 6 month intervention
  Using measured height and weight

CONTACTS AND LOCATIONS:
Overall Officials: Valarie BB Jernigan, DrPH, MPH, Principal Investigator — Oklahoma State University Center for Health Sciences; Joy Standridge, MPH, Principal Investigator — The Chickasaw Nation
Locations (1):
- The Chickasaw Nation, Ada, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No